CLINICAL TRIAL: NCT02265380
Title: A Randomized Controlled Trial to Demonstrate the Safety and Efficacy of the OptiVein IV Catheter In a Pediatric Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit patients sufficiently
Sponsor: Optomeditech Oy (Industry)
Collaborators: Hospital District of Helsinki and Uusimaa (Other); CardioMed Device Consultants, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMT-CT-002-PED
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Peripheral Venous Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment with OptiVein (Experimental): The patient will have an IV catheter placed with the use of OptiVein device.
  Interventions: Device: Placement of IV catheter
- Treatment with Vasofix Certo (Active Comparator): The patient will have an IV catheter placed with the use of Vasofix Certo device.
  Interventions: Device: Placement of IV catheter

INTERVENTIONS:
Device: Placement of IV catheter

SUMMARY:
A prospective, single-center, open-label, randomized controlled trial to demonstrate the safety and efficacy of the OptiVein IV Catheter in the pediatric population. The study hypothesis is that OptiVein IV Catheter use will be superior to the control in successful venous access after first attempt.

DETAILED DESCRIPTION:
The OptiVein System uses transillumination of skin tissue to aid in cannulation and consists of the OptiVein IV Catheter with an integrated optical fiber, and an electronic unit. The electronic unit is a portable internally powered generator of low power visible laser light of green color. The electronic unit generates visible light, which is released from the tip of the needle into the soft tissue around the tip of the IV catheter. Light is visible through the skin and helps mark the location of the tip of the needle under the skin and against the vein.

In addition to pinpointing the exact location of the tip of the needle, the OptiVein System informs the user of the exact moment of penetration of the tip of the needle into the blood vessel. Hemoglobin in blood strongly absorbs visible light of specific wavelengths, so when the needle enters the blood vessel, the light is instantly absorbed by blood, which causes instant fading of skin transillumination. Instant disappearance of tissue illumination indicates successful venipuncture. The user can then lower the angle of the needle and start to advance the cannula over the needle into the blood vessel. Such optical confirmation is much faster than the traditional observation of blood in the flashback chamber of the needle and should lead to increased first-attempt success rates and decreased cannulation-related complications.

The use of OptiVein device will be compared to the use of a traditional IV catheter to explore the potential increase of effectiveness of cannulation with OptiVein versus traditional IV catheters.

ELIGIBILITY:
Inclusion Criteria:

* Aged newborn to 12 years
* Has written or verbal order for insertion of an IV
* Requires peripheral IV therapy (catheter)
* Has an insertion site in the hand, forearm, foot, leg, or head free of deformities, phlebitis, infiltration, dermatitis, burns, lesions or tattoos
* Demonstrates cooperation with a catheter insertion and the study protocol

Exclusion Criteria:

* In the newborn nursery or intensive care units (neonatal or pediatric)
* On patient-controlled analgesia pump
* Patient is anesthetized
* Terminally ill
* Transferred from the operating room less than 8 hours postanasthesia
* Any child the research staff deem unobservable
* The study IV catheter site will be placed below an old infusion site
* The study IV site needs to be immobilized with a splint or other devices
* Has or has had a previous IV catheter related phlebitis or infiltration during current hospitalization
* Will require a power injection for a radiologic procedure during participation in this study

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 188 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-08-25 (Actual); Study Completion 2016-08-25 (Actual)

PRIMARY OUTCOMES:
Successful IV insertion on the first attempt | Immediate
  Successful IV insertion on the first attempt, defined as placement of the catheter inside the vein allowing for fluid or drug delivery or blood withdrawal.

SECONDARY OUTCOMES:
Total number of attempts required for successful IV insertion | Immediate
Time to successful IV insertion | Immediate
  Defined as time from the first skin puncture to placement of the catheter inside the vein allowing for fluid or drug delivery or blood withdrawal.
Incidence of blood extravasation resulting in a hematoma | Up to 72 hours
Incidence of fluid extravasation delivered through catheter | Up to 72 hours
Incidence of infection (phlebitis, dermatitis and induration) | Up to 72 hours
  Incidence of infection (phlebitis, dermatitis and induration) at insertion site through 72 hours or at the time of catheter removal, whichever occurs first.
Unplanned withdrawal of IV catheter | Up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tomi Taivainen, MD, PhD, Principal Investigator — Hospital District of Helsinki and Uusimaa
Locations (1):
- Helsinki and Uusimaa Hospital District, Children's Hospital, Helsinki, Finland